CLINICAL TRIAL: NCT05735197
Title: Effect of Sodium-Glucose Co-transporter 2 Inhibitors on Kidney Disease Progression and Bone Mineral Metabolism in Non-diabetic Patients With Chronic Kidney Disease
Brief Title: Effect of Dapagliflozin on Renal Outcomes and Bone Mineral Disease in Non-diabetic Chronic Kidney Disease Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mohamed Mohsen Elshayeb, Nephrology specialist at urology and nephrology center (principal investigator), Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MD.22.02.600
Record Dates: First submitted 2023-02-08; First posted 2023-02-21 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Chronic Kidney Diseases; Bone Diseases, Metabolic
Keywords: CKD; Bone mineral disease; SGLT2i
MeSH Terms: conditions — Renal Insufficiency, Chronic; Bone Diseases, Metabolic | interventions — dapagliflozin

STUDY DESIGN:
Intervention Model Description: 100 patients with non-diabetic CKD with an estimated glomerular filtration rate (eGFR) of 25-75 ml/min/1.73m2 will be randomized into two groups:
  * Study group: includes 50 patients, they will receive SGLT2i as add on drug, Dapagliflozin 10 mg will be used once daily with or without food.
  * Control group: includes 50 patients, they will receive placebo plus their medication.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dapagliflozin group (Active Comparator): Includes 50 patients, they will receive SGLT2i as add on drug, Dapagliflozin 10 mg will be used once daily with or without food.
  Interventions: Drug: Dapagliflozin 10mg Tab
- Placebo group (Placebo Comparator): Includes 50 patients, they will receive placebo plus their medication.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dapagliflozin 10mg Tab — Dapagliflozin which is (SGLT2 inhibitor) will be used as add on medication.
  Other Names: Dapagliflozin
  Arms: Dapagliflozin group
Drug: Placebo — Placebo which has the same shape as Dapagliflozin but without active ingredient will be used as add on medication for control group.
  Other Names: control
  Arms: Placebo group

SUMMARY:
It is a randomized controlled trial in which 100 non diabetic chronic kidney disease (CKD) patient is being participated.

Their estimated glomerular filtration rate (eGFR) between 25-75 ml/min/1.73 m2.

Participants will be randomized into two groups:

* Study group: includes 50 patients, they will receive Sodium glucose co-transporter 2 inhibitor (SGLT2i) as add on drug, Dapagliflozin 10 mg will be used once daily with or without food.
* Control group: includes 50 patients, they will receive placebo their medication.

The investigators will follow up all patients for 12 months and compare their results.

This study aims to:

1. Assess SGLT2i role in delaying the progression of ongoing chronic kidney disease.
2. Study the impact of SGLT2i on bone and mineral metabolism in this patients' population.

DETAILED DESCRIPTION:
All patients have been recruited from the renal clinic of Nephrology and transplantation unit. The entire study will be conducted at Urology and Nephrology center in Mansoura University.

Study design and sample size:

• Sample size: Was calculated based on previous research by (DAPA-CKD) study using G. power program with α error 0.05 and power 80% and it was equal to approximately 98 patients.

Type of the study: Randomized, controlled trial.

Patient's enrollment: 100 patients with non-diabetic CKD with an estimated glomerular filtration rate (eGFR) of 25-75 ml/min/1.73m2 will be randomized into two groups:

* Study group: includes 50 patients, they will receive SGLT2i as add on drug, Dapagliflozin 10 mg will be used once daily with or without food.
* Control group: includes 50 patients, they will receive placebo plus their medication.

The investigators will follow up all patients for 12 months and compare their results.

Study Protocol:

• 100 patients will be included in the study. Patients will be randomized 1:1, either to a control group receiving placebo and an intervention group receiving 10 mg dapagliflozin daily.

The following data will be gathered and evaluated for all patients:

I- Baseline evaluation:

* Patients of both groups will be subjected to full history taking including duration and cause of CKD and drug history and routine clinical examination.
* Laboratory investigations:

  1. Serum creatinine, calcium, phosphorus and magnesium.
  2. 24 hour urine protein, Creatinine clearance, calcium and phosphorus
  3. Urine analysis with microscopy and random urine protein/creatinine ratio.
  4. Random blood sugar.
  5. Intact parathyroid hormone (iPTH).
  6. Urine pregnancy test for females in child bearing period.
  7. Bone turnover markers:

     1. Bone-specific alkaline phosphatase (BALP).
     2. Propeptides of type I procollagen (P1NP).
     3. Carboxy-terminal crosslinked telopeptide of type 1 collagen (CTX-1).
     4. Tartrate-resistant acid phosphatase (TRAP-5b).
* Radiological investigation:

Quantitative computed tomography: to detect cortical and trabecular bone density.

II-Evaluation throughout the study:

All patients will be evaluated every 3 months thereafter regarding:

* Thorough clinical evaluation including regular measurement of blood pressure and assessment of volume status each visit.
* Laboratory investigations:

  1. Serum creatinine, calcium, phosphorus and magnesium.
  2. 24 hour urine protein, Creatinine clearance, calcium and phosphorus
  3. Urine analysis with microscopy and random urine protein/creatinine ratio.
  4. Random blood sugar.

All patients will be evaluated at 12 month regarding:

1. iPTH
2. Bone turnover markers:

   * Bone-specific alkaline phosphatase (BALP)
   * Propeptides of type I procollagen (P1NP).
   * Carboxy-terminal crosslinked telopeptide of type 1 collagen (CTX-1).
   * Tartrate-resistant acid phosphatase (TRAP-5b).
3. Quantitative computed tomography (QCT).

The main research question is: Does use of SGLT2i will slow down the progression of CKD in patients without diabetes? Will the use of SGLT2i have a negative impact on bone and mineral metabolism among these patients?

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged more than 18 year.
2. CKD patient with eGFR from 25 to 75 ml/min/1.73m2 with no evidence of acute drop of the GFR in the last 3 months.
3. Willing to sign informed consent.

Exclusion Criteria:

1. eGFR less than 25 ml/min per 1.73 m2.
2. Medical history of chronic disease (diabetes mellitus, chronic liver and/or respiratory diseases).
3. Patients with primary or secondary glomerulonephritis/ nephrotic syndrome (proteinuria ≥ 3.5 gm/day) and/or any evidence of active immunological/ collagen vascular disease.
4. Inability to sign the study consent form or refusal to participate in the study.
5. Evidence of urinary obstruction.
6. Patients with evidence of volume depletion or receiving a combination of angiotensin converting enzyme (ACE) inhibitors and angiotensin receptor blockers (ARBS)..
7. Patients with current history of frequent hypotensive episodes or systolic blood pressure <100 mmHg.
8. Patients with history of recurrent urinary tract infection and/or valvovaginitis
9. Patients with ongoing active malignancy.
10. Patients with any evidence of active infection including human immunodeficiency virus (HIV), hepatitis B virus (HBV), hepatitis C virus (HCV) and tuberculosis (TB).
11. Current or previous organ transplantation, or expected to get a kidney transplant within 12 months.
12. Patients who received any SGLT2i for more than 3 months in the past.
13. Patients who are already on medications that may affect or interact with bone metabolism such as bisphosphonates, calcitonin, steroid, denosumab and estrogen during the last 6 months.
14. Pregnant and/or lactating woman.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-08-10 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Effect of dapagliflozin on CKD progression | 1 year
  effect of Dapagliflozin on eGFR (ml/min)
Effect of dapagliflozin on Bone | 1 year
  effect on serum levels of bone turnover markers measured by ELISA
Effect of dapagliflozin on minerals | 1 year
  effect of Dapagliflozin on calcium, phosphorus and magnesium
Effect of dapagliflozin on BMD | 1 year
  assess Bone mineral disease (BMD) by using quantitative CT (QCT)

SECONDARY OUTCOMES:
Effect of dapagliflozin on blood pressure | 1 year
  follow up systolic and diastolic blood pressure throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Mohsen elshayeb, Msc, Principal Investigator — Mansoura Urology and nephrology center, Mansoura University
Locations (1):
- Urology and Nephrology center, Mansoura University, Al Mansurah, Aldakahliya, Egypt

IPD SHARING:
Plan to Share IPD: Yes
all individual participant data (IPD) that underlie results in publication
Supporting Information: Study Protocol, CSR